CLINICAL TRIAL: NCT01058343
Title: A Phase I-II, Randomized, Double-blind, Placebo-controlled, Dose Escalation Study of Neovacs' IFNα-Kinoid in Adult Subjects With Systemic Lupus Erythematosus.
Brief Title: Safety of IFNa Kinoid in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neovacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IFN-K-001
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- IFN-K 1 (Experimental): IFN kinoid dose 1
  Interventions: Biological: IFN-K
- IFN-K-2 (Experimental): IFN kinoid dose 2
  Interventions: Biological: IFN-K
- IFN-K 3 (Experimental): IFN kinoid dose 3
  Interventions: Biological: IFN-K
- IFN-K 4 (Experimental): IFN kinoid dose 4
  Interventions: Biological: IFN-K
- Saline (Placebo Comparator): saline at same dose as IFN K
  Interventions: Biological: IFN-K

INTERVENTIONS:
Biological: IFN-K — 3 to 4 IM injections over 3 months

SUMMARY:
Interferon alpha (IFNa) is involved in the pathogenesis of systemic lupus erythematosus (SLE)and IFNa levels are associated with the severity of the disease. Blocking IFNa could be an attractive therapeutic strategy. Active immunization with IFNa kinoid (IFN-K) induces a polyclonal antibody response.

This study will evaluate the safety of IFN-K in patients with mild to moderate SLE. It will also measure the induction of anti-IFNa antibodies and evaluate the clinical impact on SLE disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of SLE according to current American College of Rheumatology (ACR) criteria (4 of 11 ACR criteria),
* 2. SLEDAI ≥4 and ≤10,
* 3. Positive Anti-nuclear Antibodies (ANA) and/or Positive anti-dsDNA antibodies
* 4. Male or female between 18 and 50 years of age
* 5. Current immunity to measles, mumps, rubella and varicella, as evidenced by positive IgG titers at the time of screening,
* 6. For subjects recruited during local influenza season, current vaccination against seasonal influenza at least 7 days prior to randomization,
* 7. Vaccination against H1N1 influenza at least 7 days prior to randomization.
* 8. For subjects with reproductive potential (males and females), use of a reliable means of contraception
* 9. Written informed consent obtained from the subject.

Exclusion Criteria:

* 1. Any serious manifestation of lupus at entry, that, in the opinion of the investigator is likely to require initiation of off-protocol medication changes during the course of the study and in particular no BILAG A score,
* 2. Any non-SLE manifestation likely to require, in the investigator's judgment, treatment with high-dose corticosteroids or the addition of an immunosuppressive regimen during the course of the trial,
* 3. Received > 20 mg/day of prednisone equivalent for > 7 days during the 30 days prior to screening,
* 4. Currently receiving or having received pulse dose corticosteroids or intravenous immunoglobulin (IVIg) within 3 months prior to screening,
* 5. Received cyclophosphamide within 3 months prior to screening,
* 6. Received a monoclonal antibody during the 6 months prior to screening,
* 7. Previously received an investigational treatment directed against IFNa,
* 8. Received B-cell depleting therapy (e.g. Rituximab) within 12 months
* 9. Received IV antibiotics during the 30 days prior to screening,
* 10. Significant electrocardiogram (ECG) abnormalities ,
* 11. Evidence of any clinically significant abnormality on a chest X-ray which, in the opinion of the investigator could represent active infection, latent tuberculosis or treatable manifestation of lupus,
* 12. Any laboratory abnormality that is clinically relevant
* 13. History of malignancy except completely excised basal cell carcinoma,
* 14. Congenital immune deficiency,
* 15. Positive IgM antibody titers in the presence of negative IgG titers to Epstein-Barr virus (EBV) or cytomegalovirus (CMV),
* 16. Frequent recurrences of oral or genital herpes simplex lesions (≥ 6 / year),
* 17. Episode of shingles within one year of screening,
* 18. Human Immunodeficiency Virus (HIV), hepatitis C virus (HCV) or HBV (HBsAg, anti-HBc ab) positive,
* 19. Any current signs or symptoms of infection at entry,
* 20. Administration of any live vaccine within the 3 months prior to study entry
* 21. Planned use of any investigational or non-registered product

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | study duration

SECONDARY OUTCOMES:
Proportion of patients with anti IFNa antibodies | Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jorgensen, MD, PhD, Principal Investigator — Unité Clinique d'Immuno-Rhumatologie Thérapeutique, Hôpital Lapeyronie, Montpellier, France
Locations (14):
- Cliniques Universitaires St Luc, Brussels, Belgium
- MHAT "Sveti Ivan Rilski", Sofia, Bulgaria
- Croatia (2):
  - University Hospital Split, Split
  - KBC Zagreb, Zagreb
- France (5):
  - Hopital Claude Huriez, Lille
  - Hopital Lapeyronie, Montpellier
  - Hopital de la Pitie Salpetriere, Paris
  - Hopital du Kremlin Bicetre, Paris
  - Hopital Haut-Leveque, Pessac
- Germany (2):
  - Kerckhoff-Klinik Gmbh, Bad Nauheim
  - Charite, Berlin
- Switzerland (3):
  - Inselspital, Bern
  - Geneva University Hospital, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Derived] Ducreux J, Houssiau FA, Vandepapeliere P, Jorgensen C, Lazaro E, Spertini F, Colaone F, Roucairol C, Laborie M, Croughs T, Grouard-Vogel G, Lauwerys BR. Interferon alpha kinoid induces neutralizing anti-interferon alpha antibodies that decrease the expression of interferon-induced and B cell activation associated transcripts: analysis of extended follow-up data from the interferon alpha kinoid phase I/II study. Rheumatology (Oxford). 2016 Oct;55(10):1901-5. doi: 10.1093/rheumatology/kew262. Epub 2016 Jun 28. PMID 27354683
- [Derived] Lauwerys BR, Hachulla E, Spertini F, Lazaro E, Jorgensen C, Mariette X, Haelterman E, Grouard-Vogel G, Fanget B, Dhellin O, Vandepapeliere P, Houssiau FA. Down-regulation of interferon signature in systemic lupus erythematosus patients by active immunization with interferon alpha-kinoid. Arthritis Rheum. 2013 Feb;65(2):447-56. doi: 10.1002/art.37785. PMID 23203821